Laureate Institute for Brain Research, Inc., Tulsa, OK, United States

| RESEARCH SUBJECT INFORMATION AND CONSENT FORM – PHASE 2 | |
|---|---|
| TITLE: | Developing and Evaluating a Positive Valence Treatment for |
| | Alcohol Use Disorder with Anxiety or Depression |

This consent form contains important information to help you decide whether to participate in a research study.

The study staff will explain this study to you. Ask questions about anything that is not clear at any time. You may take home an unsigned copy of this consent form to think about and discuss with family or friends.

- > Being in a study is voluntary your choice.
- > If you join this study, you can still stop at any time.
- > No one can promise that a study will help you.
- > Do not join this study unless all of your questions are answered.

# After reading and discussing the information in this consent form you should know:

- Why this research study is being done;
- What will happen during the study;
- Any possible benefits to you;
- The possible risks to you;
- Other options you could choose instead of being in this study;
- How your personal health information will be treated during the study and after the study is over;
- Whether being in this study could involve any cost to you; and
- What to do if you have problems or questions about this study.

## Please read this consent form carefully.

#### RESEARCH SUBJECT INFORMATION AND CONSENT FORM - Phase 2

TITLE: Developing and Evaluating a Positive Valence Treatment for

Alcohol Use Disorder with Anxiety or Depression

**PROTOCOL NO.:** 2022-003

WCG IRB Protocol #20223794

2022-003

**SPONSOR:** Laureate Institute for Brain Research (LIBR)

**INVESTIGATOR:** Robin Aupperle, PhD

6655 S Yale Ave

Tulsa, Oklahoma 74136

**United States** 

STUDY-RELATED

PHONE NUMBER(S): Robin Aupperle, PhD

918-502-5744

918-481-4000 (24 hours)

Samantha Ramirez

918-859-1708

## RESEARCH CONSENT SUMMARY

You are being asked for your consent to take part in a research study. This document provides a concise summary of this research. It describes the key information that we believe most people need to decide whether to take part in this research. Later sections of this document will provide all relevant details.

#### What should I know about this research?

Someone will explain this research to you.

Taking part in this research is voluntary. Whether you take part is up to you.

If you don't take part, it won't be held against you.

You can take part now and later drop out, and it won't be held against you If you don't understand, ask questions.

Ask all the questions you want before you decide.

#### How long will I be in this research?

We expect that your taking part in this research will last about 18-24 weeks.

#### Why is this research being done?

The purpose of this research is to study the effects of an investigational intervention focusing on positivity (affective modulation of positivity, AMP) compared to an intervention focusing on the connection between thoughts, emotions, and behaviors (cognitive behavioral therapy, CBT) on those with comorbid anxiety or depression and alcohol use disorder.

## What happens to me if I agree to take part in this research?

If you decide to take part in this research study, the general procedures include attending treatment sessions in the clinic, answering questionnaires and surveys, and having MRIs.

## Could being in this research hurt me?

The most important risks or discomforts that you may expect from taking part in this research include feeling uncomfortable from the questions asked, worsening mental health or substance use symptoms or behaviors, having feelings of claustrophobia and anxiety from the MRI, and loss of confidentiality.

## Will being in this research benefit me?

The most important benefits that you may expect from taking part in this research include a decrease in symptoms or increase in positive emotions, although this cannot be guaranteed. Possible benefits to others include learning more about the potential of interventions focusing on positivity.

## What other choices do I have besides taking part in this research?

Instead of being in this research, your choices may include other options to obtain therapy for anxiety/depression, alcohol use disorder, or other symptoms and conditions you may be experiencing like approved medications and/or different talk therapies.

## **DETAILED CONSENT**

Taking part in this research is voluntary. You may decide not to participate, or you may leave the study at any time. Your decision will not result in any penalty or loss of benefits to which you are otherwise entitled.

If you have any questions, concerns, or complaints or think this research has hurt you, talk to the research team at the phone number(s) listed in this document.

This consent form describes a research study. Research studies involve only individuals who choose to participate. Please take your time to make your decision about participating in the study.

This consent form may contain words that you do not understand. Please ask the Principal Investigator or the study staff to explain any words or information that you do not clearly understand. You may take home an unsigned copy of this consent form to think about or discuss with family or friends before making your decision.

## Why Have You Been Asked To Participate In This Study?

You are being asked to take part in this study because:

 You have reported symptoms associated with alcohol use disorder AND you have reported symptoms associated with anxiety or depression

## Why Is This Study Being Done?

This project seeks to study the effects of an investigational intervention focusing on enhancing positive emotions (affective modulation of positivity, AMP) compared to an intervention focusing on the connection between thoughts, emotions and behaviors (cognitive behavioral therapy, CBT) on anxiety or depression and alcohol use.

## What Devices Are Involved In This Study?

Magnetic Resonance Imaging (MRI – use of a magnetic field to produce an image) is used in this study to look at brain function and anatomy. A physiological recording system will also be used to monitor bodily sensations, such as heart rate and breathing.

## **How Many Subjects Will Take Part In The Study?**

About 100 subjects will take part in this study at the Laureate Institute for Brain Research.

## What Is Involved In The Study?

If you take part in this study, you may have the following tests and procedures at the Laureate Institute for Brain Research (LIBR):

## Interview & Questionnaires

You will be asked to complete questionnaires. These questionnaires will ask about your health and substance use behaviors and mental and physical states. You will have an interview with a member of the research staff. You will be asked will be asked a series of questions about your mental and physical health, substance abuse and symptoms, and important events you may have experienced during your lifetime. This part of the visit will last about 1.5 - 3 hours. We may ask permission to audio record portions of the interviews and assessments for study purposes only.

## <u>Urine Drug Tests and Breathalyzer</u>

You will be asked to complete urine drug tests at the pre- and post-treatment sessions and the 3 month follow-up visit, as well as alcohol breathalyzer tests repeatedly throughout the study.

#### Magnetic Resonance Imaging (MRI)

For MRI studies, you will be given a brief medical history questionnaire and screening form to complete. Undesirable medical findings may arise during the interview, screening, or MRI scanning. If so, these findings will remain confidential and will be discussed with you by a researcher of this study.

Before MRI scanning, you will learn tasks that will involve (a) responding to positive and negative emotional images and sounds, (b) making decisions when faced with potential emotional or rewarding outcomes. Training for the MRI tasks will last approximately 15 minutes. You will then be placed in the MRI scanner to perform the tasks. The MRI scanner rapidly takes pictures of your brain. The MRI scanner is a metal tube surrounded by a strong magnetic field. During the MRI, you will lie on a table that can slide in and out of the tube. You will be asked to lie still during scanning. Earplugs will be provided to lessen the loud "knocking" sounds that the scanner makes while it is imaging your brain.

First, you will receive a series of short scans that allow us to know where your head is inside the tube. You will then receive a scan lasting 5 to 15 minutes that gives us more detailed pictures of your brain. Finally, you will undergo a series of scans lasting about 50 minutes during which you will perform the tasks and or look at a cross on the screen. During all of these scans, it will be very important to remain still. Your time in the scanner will be about 1.5 hours.

If you are a female, a urine pregnancy test will be obtained. An over-the-counter urine pregnancy test will be completed just prior to any MRI scanning. You will not be allowed to participate in the study if the pregnancy test reads positive.

## **Treatment**

You will be randomly assigned to AMP or CBT treatment, meaning you will have a 1 in 2 chance of being in either group. You will come into the clinic once or twice per week for 12 treatment sessions. Each session will last about 1 - 1.5 hours.

If you are in the AMP group, during each session you will be presented with educational materials and prescribed exercises designed to increase positive thoughts, behaviors, and emotions. Use of alcohol will be discussed within the context of the intervention.

If you are in the CBT group, during the sessions you will be presented with educational materials and prescribed exercises designed to increase your awareness of how thoughts, emotions, and behaviors relate to one another – particular as they are relevant to alcohol use.

You will also be given instructions for completing activities throughout the week based on the information provided each session, including rating forms to assess your emotions and reactions to the exercises. These sessions will be video or audio recorded to make sure that the treatment protocol is being administered the same way to each participant. You will be asked to complete brief surveys at each intervention session, related to your mental health.

In addition to the in-person therapy sessions, you will be provided between-session assignments to complete as part of that therapy. You may also be contacted by clinicians or research staff in between sessions for scheduling purposes or to check in regarding therapy assignments.

All therapy sessions will be led by a licensed Clinical Social Worker, licensed Clinical Psychologist, or a psychologist or therapist in training (e.g., individuals working towards clinical master's or doctoral degree or license). Each therapy session will be video and/or audio recorded and may be reviewed by the research team and/or affiliated consultants that are experts in the therapy being provided. The recordings may be used for educational and training purposes of clinical staff that may or may not be affiliated with LIBR. The recording(s) may include your first name, and partial or full facial pictures. The recording(s) will be stored at LIBR on secure servers that are password protected. Recordings will be identified by therapy session name and will not include identifiable information of individual participants. Recordings will be retained indefinitely for training and supervisory purposes.

Individual treatment sessions may be conducted virtually utilizing video conferencing technology. Depending upon your preference, you and the therapist may also communicate using email, text, or voice messages. We cannot guarantee confidentiality of information shared during videoconferencing or phone- or email-based communication methods.

## How Long Will You Be In The Study?

There will be 1-2 baseline visits lasting approximately 3-4 hours long total, after which there will be 12 therapy sessions completed within 14 weeks, each lasting approximately 1 - 1.5 hours each. After completing these sessions, there would be 1-2 post-treatment sessions lasting approximately 2-3 hours total. Additionally, there will be a follow up visit approximately 3 months after your last treatment session that will also take approximately 2-3 hours total.

For those who opt to complete the brain imaging part of the study, this will involve an additional session at baseline and an additional session after treatment, each of which will last approximately 3 hours.

There may be circumstances under which your participation in the study may be stopped by the investigator without your consent; for example, if it is identified via one of the assessments that you do not meet criteria for the study. There may also be times in which completion of the intervention involved in the study is considered not in your best interest, such as if you experience physical or mental health symptoms requiring immediate medical attention. Under these circumstances, your participation may be stopped without your consent.

You may stop participating in this study at any time.

## What Are The Risks Of The Study?

The study may involve the risks described in this section.

It is possible that your participation in this study might reveal unanticipated medical or psychiatric findings. You have the right to refuse to answer any question that you do not wish to answer and to withdraw from participating in the study at any time.

This study is being done to determine the potential benefit of interventions for individuals experiencing alcohol use disorder and symptoms of depression or anxiety. The interventions involved in the study has been found beneficial for individuals experiencing mood and/or anxiety symptoms in previous research but have not been as fully studied in relation to alcohol use disorder. It is possible that medical or psychiatric problems may arise or be identified during the screening process, for which we may not be able to provide therapy. It is important that you understand that therapy for medical or psychiatric conditions other than mild to moderate depression and/or anxiety and alcohol use disorder will not be offered in this study.

If unanticipated findings occur, we will provide you with all results of screening tests and will assist you in communicating these results to your primary physician or other health care provider, so long as you provide written consent for us to do so.

There is risk of loss of confidentiality.

The risks of the study procedures are listed and discussed below.

## Risks Associated with Interview, Questionnaires, and Behavioral Testing

The interview and questionnaires about your health, mood, and behavior are not physically harmful but may be stressful to complete. We ask only that you try your best. You may stop any test at any time. In particular, the behavioral tests may include negative or triggering images, such as those associated with alcohol use. We ask that you try your best and inform study staff of significant distress or increases in symptoms or alcohol craving that you may experience. It is possible that being asked personal questions about your emotions and mood, personality, and behavior may make you feel uncomfortable. You may skip questions that make you feel uncomfortable.

## Risks of MRI scanning

People are at risk for injury from the MRI magnet if they have any of the following metal implants or fragments:

- pacemakers or other implanted electronic devices
- brain stimulators
- dental implants
- aneurysm clips (metal clips on the wall of a large artery)
- metallic prostheses (including metal pins and rods, heart valves, and cochlear implants)
- permanent eyeliner
- implanted delivery pump
- shrapnel fragments

You will be asked to complete an MRI screening form for the MRI scan. You will be screened for these implants or metal fragments before the study, and if you have any of

them, you will not receive an MRI scan and cannot be in the study. Tell the study doctor if you are uncertain whether you have any metal objects in your body. In addition, all magnetic objects (for example, watches, coins, jewelry, and credit cards) must be removed before entering the MRI scanner room.

Welders and metal workers are also at risk for injury because they may be unaware of small metal fragments in the eye.

There are no known long-term risks or consequences of MRI scans. However, you may become uncomfortable because you will be lying in a small space. Some people are bothered by the loud thumping noises made by the scanner. You will wear earplugs to reduce the noise and increase your comfort during scanning. LIBR study staff will closely and continuously monitor you throughout the scanning procedure. You will be able to use an emergency call button at all times during the scan. You will be removed from the scanner immediately if you request to be removed.

If you are a female, it is best that you not be pregnant while participating in this study. A urine-based pregnancy test may be obtained prior to any MRI scanning.

## Risks associated with treatment:

It is possible that you may experience adverse effects to treatment in the form of worsening mental health or substance use symptoms or behaviors. You will be monitored weekly for a change in your symptoms by researchers. A clinical psychologist and psychiatrist are part of the research team.

## Are There Benefits To Taking Part In The Study?

There may or may not be any direct benefit to you from participating in this study. All subjects in the study will be receiving treatment and it is possible that you may experience a decrease in symptoms or increase in positive emotions as a result of these procedures. However, benefit from the treatment cannot be guaranteed.

## What Are The Costs Of Participating In The Study?

Neither you nor your health insurance will be charged for any of the study tests, procedures, or activities. If you need to be hospitalized, voluntarily or involuntarily, Laureate Institute for Brain Research does not intend to provide payment for this, and you or your insurance provider will be billed for these costs.

## Will You Be Paid For Participating In This Study?

For pre- and post- treatment sessions, you will be paid \$10 per half hour for completion of the interview and questionnaires. While you are prepped for MRI scanner and while in the MRI scanner, you will be paid \$25 per half hour. Your time in the MRI scanner will be approximately 1 ½ hours. You may earn up to \$55 more based on your participation in the decision-making tasks.

For assessments completed at the intervention sessions, you will be compensated \$5 per session. No compensation will be provided for procedures associated with the intervention itself.

You will be paid through a ClinCard (similar to a debit card) that may be used 24 hours after the visit.

## What Other Options Are There?

This study is for research purposes only, so your other option is not to participate in the study.

While the therapies being provided as part of this study have been found to be beneficial for individuals experiencing depression and/or anxiety, there are other options to obtain therapy for these symptoms, alcohol use disorder, or other symptoms and conditions you may be experiencing. Your options may include approved medications, as well as different talk therapies than is used in the current study. Information concerning community clinics and treatment resources will be provided to you as requested.

## Confidentiality

## What information may be used and given to others?

The study doctor will get your personal and medical information which may include research records, logs about phone calls made as part of this research, and records about your study visits.

## Who may use and give out information about you?

The study investigator, study staff, and consultants.

## Who might get this information?

 Your information may be given to the study Sponsors, the Department of Health and Human Services (DHHS) agencies, and the WCG IRB. Sponsor means any persons or companies that are working for or with the sponsor, or owned by the sponsor, who is financially supporting the conduction of the research.

## Why will this information be used and/or given to others?

This information will be used and/or give to others to do the research, to study the results, and to make sure that the research was done right. If the results of this study are made public, information that identifies you will not be used.

## **Secondary Research**

There is a possibility that identifiers might be removed from the identifiable
private information or identifiable biospecimens, and after such removal, the
information or biospecimens may be used for future research studies or
distributed to another investigator for future research studies without additional
informed consent.

## **National Institute Data Archive (NDA)**

- Data from this study will be submitted to the National Institute of Mental Health's data archive, a large database where deidentified study data is stored and managed.
- Deidentified study data means that all personal information (such as name, address, birthdate and phone number) will be removed and replaced with a code number.
- Once uploaded, other researchers can request your deidentified study data.
   Every researcher (and institutions to which they belong) who requests your deidentified study data must promise to keep your data safe and promise not to try to learn your identity. Experts at the NIH who know how to keep your data safe will review each request carefully to reduce risks to your privacy.
- Sharing your study data does have some risks, although these risks are rare.
   Your study data could be accidentally shared with an unauthorized person who may attempt to learn your identity. The study researchers will make every attempt to protect your identity.
- You may not benefit directly from allowing your study data to be shared with NDA. However, study data may help researchers around the world to better understand mental health.
- You may decide now or later that you do not want your study data to be added to the NDA. You can still participate in this research study even if you decide that you do not want your data to be added to the NDA. To opt out, please provide the study staff with a written letter requesting that your data not be submitted to the NDA database.
- Once your data is part of the NDA, the study researchers cannot take back the study data that was shared before they were notified that you changed your mind. If you would like more information about NDA, this is available on-line at http://nda.nih.gov.

## What if I decide not to give permission to use and give out my health information?

Then you will not be able to be in this research study.

## May I review or copy my information?

Yes, but only after the research is over.

## May I withdraw or revoke (cancel) my permission?

Yes, but this permission will not stop automatically.

You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the study doctor. If you withdraw your permission, you will not be able to stay in this study.

When you withdraw your permission, no new health information identifying you will be gathered after that date. Information that has already been gathered may still be used and given to others.

## Is my health information protected after it has been given to others?

The information you provide as part of this study will be kept confidential within Laureate Institute for Brain Research, within the limits of the law and with the exception of therapy audio or video tapes used for supervision or training purposes. However, there is always a risk that your information will be given to others without your permission and may no longer be protected.

If you have any questions or concerns about your privacy rights, you should contact the LIBR Privacy Officer at 918-502-5155 or via email at privacy@laureateinstitute.org.

You have the right to access the medical information that has been collected about you as a part of this research study. However, you may not have access to this medical information until the entire research study is finished.

## **Certificate of Confidentiality**

We will do everything we can to keep others from learning about your participation in this study. To further help us protect your privacy, we have obtained a Certificate of Confidentiality from the United States Department of Health and Human Services (DHHS). With this Certificate, we cannot be forced (for example by court order or subpoena) to disclose information that may identify you in any federal, state, local, civil, criminal, legislative, administrative, or other proceedings. The researchers will use the Certificate to resist any demands for information that would identify you, except to prevent serious harm to you or others, and as explained below.

You should understand that a Certificate of Confidentiality does not prevent you, or a member of your family, from voluntarily releasing information about yourself, or your involvement in this study.

If an insurer or employer learns about your participation, and obtains your consent to receive research information, then we may not use the Certificate of Confidentiality to withhold this information. This means that you and your family must also actively protect your own privacy. Disclosure will be necessary, however, upon request of DHHS for the purpose of audit or evaluation, and is limited only to DHHS employees involved in the review.

Finally, you should know the research team can take steps, such as telling authorities (for example, the Police) if 1) you tell us of plans to really hurt yourself, 2) you tell us of plans to really hurt another person, or 3) we learn that a child or elder has been or is being abused or neglected.

## What If You Are Injured While Participating In This Study?

If you get hurt or sick from participating in this study, emergency medical treatment is available. In an emergency, call 911. Be sure to tell the emergency staff and other healthcare providers of your participation in this study. Contact Robin Aupperle, PhD as soon as possible at 918-502-5744 or 918-481-4000 (24 hours) if you think you have a research-related injury or illness. You or your health insurance provider will be billed to cover the cost of the medical or emergency services provided. No funds have been set aside by the Laureate Institute for Brain Research to compensate you if you are hurt or get sick. However, you still have the right to bring a lawsuit if you think you were harmed and deserve compensation.

You do not give up any of your legal rights by signing this consent form.

## Who Will Provide Funding For The Study?

Funding for this research study will be provided by Laureate Institute for Brain Research and the National Institute on Alcohol Abuse and Alcoholism.

## What Are Your Rights As A Participant?

Taking part in this study is voluntary. You may choose not to participate. Refusal to participate will involve no penalty or loss of benefits to which you are otherwise entitled. If you agree to participate and then decide against it, you can withdraw for any reason and leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

Your participation in this study may be stopped at any time by the study doctor or the sponsor without your consent for any reason, including if it is in your best interest or if you do not consent to continue in the study after being told of changes in the research that may affect you.

## What If There Are New Findings?

We will provide you with any significant new findings developed during the research study that may affect your health, welfare, or willingness to continue your participation in this study.

#### Who Should You Call If You Have Questions Or Problems?

Your contact person for this study is Samantha Ramirez. She can be reached during business hours at 918-859-1708.

IRB APPROVED Jul 29, 2022

If you have questions, about your participation in this study, concerns, or complaints about the study, or have a research-related injury, contact the study investigator, Robin Aupperle, PhD, at 918-502-5744 or 918-481-4000 (24 hours). For emergencies, call 911.

If you have questions about your rights as a research subject or if you have questions, concerns, input, or complaints about the research, you may contact:

WCG IRB

Telephone: 855-818-2289

E-mail: researchquestions@wcgirb.com

WCG IRB is a group of people who perform independent review of research. WCG IRB will not be able to answer some study-specific questions, such as questions about appointment times. However, you may contact WCG IRB if the research staff cannot be reached or if you wish to talk to someone other than the research staff.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

Do not sign this consent form unless you have had a chance to ask questions and have received satisfactory answers to all of your questions.

If you agree to be in this study, you will be given a signed and dated copy of this consent form.

IRB APPROVED Jul 29, 2022

## **Signature**

I have read the information in this consent form. I have been given an opportunity to ask questions. All my questions about the study and my participation in it have been answered.

## I Agree To Participate In This Study

I authorize the use and disclosure of my health information to the parties listed in the authorization section of this consent for the purposes described above.

| PRINTED NAME OF PARTICIPANT | |
|------------------------------------------------------------|------|
| Consent Signature | |
| PARTICIPANT SIGNATURE (18 years and older) | Date |
| SIGNATURE OF PERSON CONDUCTING INFORMED CONSENT DISCUSSION | Date |